CLINICAL TRIAL: NCT06796127
Title: Beijing Anzhen Hospital
Brief Title: A Multicenter Study of Artificial Intelligence Model for Fetal Congenital Heart Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: FCHD-MCS-02
Record Dates: First submitted 2025-01-20; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Congenital Heart Disease (CHD); Artificial Intelligence (AI)
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study addresses congenital heart disease in fetuses, a specific birth defect, by collaborating with multicenter medical institutions across China. It prospectively collects echocardiographic screening, diagnostic images, and structured parameter data from both normal and abnormal fetuses. Cases are followed up, and artificial intelligence (AI) models are developed to extract fetal heart echocardiographic image features and analyze the data. This process allows for the analysis of the AI models' accuracy, sensitivity, and specificity, and verifies the application value of AI models in fetal heart echocardiographic screening and diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Single or multiple pregnancy;
* Gestational age 16-40 weeks;
* Fetal echocardiographic images are clear and complete;
* Clinical data are complete and detailed;
* Sign informed consent and be able to cooperate with follow-up

Exclusion Criteria:

* Fetal echocardiographic images are incomplete or of poor quality that cannot be used for research;
* Refusal or loss of follow-up

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population was from 20 multi-center medical institutions in China, and pregnant women who underwent fetal echocardiography between 16 and 40 weeks of gestation.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic efficiency of AI model for fetal CHD | From enrollment to diagnostic verification, the evaluation period should not exceed 12 month.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Anzhen Hospital affiliated to Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol